CLINICAL TRIAL: NCT05871034
Title: Changes of Electrophysiology and Optical Coherence Tomography Angiography in Primary Open Angle Glaucoma After Phacoemulsification
Brief Title: Electroretinogram and Retinal Vascular Changes After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shorouq Abdelrahman Hassan, Assistant lecturer, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SAHASSAN
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Primary Open Angle Glaucoma
Keywords: OCTA: optical coherence tomography angiography; ERG: electroretinogram; POAG: primary open Angle glaucoma; V/A: visual acuity; IOP: intra ocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Control group who have cataract without Open Angle glaucoma Will under go phacoemulsification cataract surgery
  Interventions: Procedure: phacoemulsification
- Open Angle glaucoma group (Other): patients who have cataract and Open Angle glaucoma Will undergo phacoemulsification cataract surgery
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification — cataract extraction

SUMMARY:
To compare electrophysiological and Optical coherence tomography angiography of optic disc and macula changes after uneventful phacoemulsification between normal and cataractus patients with primary open angle glaucoma.

DETAILED DESCRIPTION:
* Study design: A prospective, non randomized, interventional, comparative study, control based study.
* Location: Ophthalmology department, Sohag university hospital. In this prospective study, aiming to investigate Optical coherence tomography angiography and electrophysiological changes after cataract surgery in normal and patients with POAG with cataract 1 day before operation, 1 week and 3 months postoperatively.
* Methodology The study will include 50 patients with primary open angle glaucoma associated with cataract and 50 patients have cataract without glaucoma.

Preoperative and postoperative evaluation:

All patients will be subjected to the following:

* History taking including age, gender, family history, systemic diseases, previous medications or ophthalmic surgery.
* Detailed ophthalmological examination including: Uncorrected visual acuity (UCVA), best corrected visual acuity (BCVA) by Snellen's fraction and converted into logarithm of the minimal angle of resolution LogMAR, refraction, keratometry, slit lamp biomicroscopy for anterior segment, IOP measurement by applanation tonometer, and posterior segment (Fundus) examination.
* Examination of the angle of anterior chamber by goniolens.
* OCTA disc and macula
* Pattern ERG and multifocal ERG

Surgical techniques:

Patients will be subdivided into two groups:

Group (A): normal Patients will undergo standard phacoemulsification surgery. Group (B): Patients with POAG will undergo standard phacoemulsification surgery.

* phaco technology by using (WHITESTAR SIGNATURE PRO, Abbott, USA)

* OCT angiography will be done by (Optovue, Inc., Fremont, California, USA).
* Electrophysiology will be done by (Roland consult Retimap, Germany)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged: 45-65 years old with cataract density doesn't interfere with Pre-operative imaging (N1-N2).
* Patients with primary open angle diagnosed for at least 2 years with glaucoma treatment associated with cataract (N1-N2).

Exclusion criteria:

s▪ patient with PACG.

* Previous intraocular surgery.
* Associated ocular or intra ocular inflammation
* Previous history of eye trauma.
* Associated intraocular pathology

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pattern and multifocal electroretinogram and Optical coherence tomography angiography of optic disc and macula changes after phacoemulsification in primary open angle glaucoma | before operation and 1st month, 3rd month post operative
  electrophysiology and optical coherence tomography angiography changes

SECONDARY OUTCOMES:
Visual acuity and intra ocular pressure changes | before operation and 1st month, 3rd month post operative
  visual acuity and intraocular pressure changes

CONTACTS AND LOCATIONS:
Overall Officials: shorouq abdelrahman, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No